CLINICAL TRIAL: NCT06059963
Title: A Prospective, Multi-center, Observational Study for Signal-C Test Evaluation
Status: Recruiting | Type: Observational
Sponsor: Universal Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: CRC-US-003
Record Dates: First submitted 2023-09-20; First posted 2023-09-29 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; Advanced Adenocarcinoma
Keywords: Advanced Precancerous Lesions
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood sample collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Average risk: Patients aged between 45 and 84, who are at average risk of developing colorectal cancer, and are scheduled for a standard-of-care screening colonoscopy.
  Interventions: Device: Signal-C™

INTERVENTIONS:
Device: Signal-C™ — Signal-C™ is a qualitative next generation sequencing-based in vitro diagnostic assay that uses targeted hybridization-based capture next-generation sequencing together with bioinformatics and machine learning algorithm for detection and combination of methylation and fragmentation associated DNA marker regions. Signal-C™ utilizes circulating cell-free DNA (cfDNA) isolated from plasma of peripheral whole blood collected via venipuncture in Streck Cell-Free DNA Blood Collection Tubes (BCTs).

SUMMARY:
To evaluate the performance characteristics of Signal-C™ a plasma circulating free-DNA test, to detect colorectal cancer and advanced precancerous lesions (APL) in an average risk screening population for 45 and over.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 45-84 years at time of consent
2. Intended to undergo a standard-of-care screening colonoscopy
3. Considered by a physician or healthcare provider as being of 'average risk' for CRC
4. Willing to consent to blood draw prior to bowel preparatory procedures or undergoing colonoscopy ideally within 90 days of the date of the investigational blood draw.
5. Willing to consent to follow-up for one year as per protocol
6. Able and willing to sign informed consent

Exclusion Criteria:

1. Undergoing colonoscopy for investigation of CRC risk symptoms
2. Has undergone colonoscopy within preceding 9 years
3. Positive FIT/FOBT result within the previous 12 months (+/- 3 months)
4. Has completed Cologuard or Epi proColon testing within the previous 3 years.
5. Has undergone a CT colonography in the prior 4 years.
6. History of colorectal cancer.
7. History of any malignancy within prior 5 years.
8. Known diagnosis of inflammatory bowel disease (IBD), including chronic ulcerative colitis (CUC) and Crohn's disease (CD).
9. Positive family history of colorectal cancer, defined as having a first- degree relative (parent, sibling, or child) with CRC diagnosed at age <60 years or with more than one first-degree relative diagnosed with CRC at any age.
10. Known hereditary/germline risk of colorectal cancer (for example, Lynch syndrome or Hereditary Non-Polyposis CRC [HNPCC], or Familial Adenomatous Polyposis [FAP]).
11. Any major physical trauma (e.g., disruption of tissue, surgery, organ transplant, blood product transfusion) within the 30 days leading up to the provision of informed consent.
12. Known medical condition which, in the opinion of the investigator, should preclude enrollment into the study.
13. Known pregnancy at informed consent, blood sample collection, and during study participation.
14. Participation in a clinical research study in which an experimental medication has been administered or may be administered within the 30 days leading up to providing informed consent or may be administered through the time of colonoscopy.

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged between 45 and 84, who are at average risk of developing colorectal cancer, and are scheduled for a standard-of-care screening colonoscopy.
  Approximately 12,000 subjects will need to be enrolled. Enrollment is event-driven and will be stopped when the required number of CRC cases have been confirmed with a final histopathological diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 1 year
  The primary objective of this study is to determine the sensitivity for CRC and specificity for advanced neoplasia (AN). Advance Neoplasia (AN) is defined as a final diagnosis of CRC or Advanced Precancerous Lesion (APL).

SECONDARY OUTCOMES:
Secondary Objective | 1 year
  To determine sensitivity for advanced precancerous lesions (APL). To determine NPV and PPV for colorectal cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Consultants of SW Virginia, Raonoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No